CLINICAL TRIAL: NCT02920970
Title: The Clinical Comparison of Narafilcon A and Stenfilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-71 (C16-601)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- narafilcon A (Active Comparator): Participants are randomized to wear narafilcon A lens pair for one week during the cross over study.
  Interventions: Device: narafilcon A
- stenfilcon A (Active Comparator): Participants are randomized to wear stenfilcon A lens pair for one week during the cross over study.
  Interventions: Device: stenfilcon A

INTERVENTIONS:
Device: narafilcon A — contact lens
  Arms: narafilcon A
Device: stenfilcon A — contact lens
  Arms: stenfilcon A

SUMMARY:
This study aims to compare the clinical performance and subjective acceptance of the narafilcon A lens with the stenfilcon A lens when used on a daily wear, daily disposable basis.

DETAILED DESCRIPTION:
This will be a randomized, subject-masked, crossover, bilateral study, controlled by cross comparison. Seventy subjects will use each lens type for a week in a random sequence. Follow-up visits for each lens will be performed after one week of wear. Lenses will be worn on a daily wear, daily disposable wear schedule.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They are of legal age (18) and capacity to volunteer.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research for the duration of this study.
  5. They have a contact lens spherical prescription between -1.00 to - 6.00D (Diopters) (inclusive)
  6. They have a spectacle cylindrical correction of -0.75D or less in each eye.
  7. They can be satisfactorily fitted with the study lens types.
  8. At dispensing, they can attain at least 0.10 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
  9. They currently use soft contact lenses or have done so in the previous six months.
  10. They are willing to comply with the wear schedule (at least six days per week and for at least eight hours per day).
  11. They own a wearable pair of spectacles.

Exclusion Criteria:

* Subjects will not be eligible to take part in the study if:

  1. They have an ocular disorder which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They have had cataract surgery.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  7. They are pregnant or breast-feeding.
  8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
  9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
  10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.
  11. They currently wear either the stenfilcon A lens or narafilcon A lens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, FAAO, FBCLA, Study Director — Eurolens Research, University of Manchester
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 72 participants were enrolled in the study, of which 70 were dispensed a contact lens to wear and 2 failed screening.
Groups:
- Stenfilcon A First Then Narafilcon A: Participants are randomized to wear stenfilcon A lens first for one week then narafilcon A.
- Narafilcon A First Then Stenfilcon A: Participants are randomized to wear narafilcon A lens first for one week then stenfilcon A.
Period: First Intervention
Arm/Group | Stenfilcon A First Then Narafilcon A | Narafilcon A First Then Stenfilcon A
Started | 38 | 32
Completed | 38 | 30
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention
Arm/Group | Stenfilcon A First Then Narafilcon A | Narafilcon A First Then Stenfilcon A
Started | 38 | 30
Completed | 37 | 30
Not Completed | 1 | 0
Not completed — Poor Lens Fit | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Number of Baseline Participants: Total number of participants enrolled in the study.
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Ocular Physiology
Description: Ocular physiology assessment of narafilcon A and stenfilcon A lenses by biomicroscopy (Scale 0-4, 0.25 steps, 0=normal, 4=severe).
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A due to protocol deviations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
units on a scale
  Conjuctival hyperaemia | 0.84 (0.25) | 0.76 (0.27)
  Limbal hyperaemia | 0.75 (0.28) | 0.62 (0.31)
  Corneal vascularisation | 0.05 (0.14) | 0.03 (0.09)
  Microcysts | 0.00 (0.00) | 0.00 (0.00)
  Oedema | 0.00 (0.00) | 0.00 (0.00)
  Corneal staining | 0.31 (0.41) | 0.33 (0.40)
  Conjuctival staining | 0.57 (0.49) | 0.76 (0.64)
  Papillary conjuctivitis | 1.01 (0.35) | 1.00 (0.31)

2. Primary Outcome: Visual Acuity
Description: Visual acuity for narafilcon A and stenfilcon A are assessed by LogMAR. High contrast is measured with black letters on a white background. Low contrast is measured with gray letters on a white background.
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at follow up due to protocol deviations.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Stenfilcon A: Participants are randomized to wear stenfilcon A lens pair and assessed after one week during the cross over study.
- Narafilcon A: Participants are randomized to wear narafilcon A lens pair and assessed after one week during the cross over study.
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
LogMAR
  High Contrast | -0.12 (0.07) | -0.10 (0.08)
  Low Contrast | 0.17 (0.09) | 0.17 (0.10)

3. Primary Outcome: Comfort Level of Stenfilcon A and Narafilcon A Lenses
Description: Subjective responses for overall comfort will be evaluated for each pair using questionnaire (Scale 0-100, 0=causes pain, cannot be tolerated, 100=excellent, cannot be felt).
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
units on a scale | 91.4 (9.8) | 83.1 (14.8)

4. Primary Outcome: Dryness of Stenfilcon A and Narafilcon A Lenses
Description: Subjective responses for dryness will be evaluated for each pair using questionnaire (Scale 0-100, 0=extremely poor, high levels of dryness, 100=excellent, no dryness).
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A due to protocol deviations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
units on a scale | 82.1 (17.2) | 81.2 (16.7)

5. Primary Outcome: Vision of Stenfilcon A and Narafilcon A Lenses
Description: Subjective responses for vision will be evaluated for each pair using questionnaire (Scale 0-100, 0=unacceptable, lens cannot be worn, 100=excellent).
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
units on a scale | 91.4 (9.4) | 88.4 (14.6)

6. Primary Outcome: Lens Surface - Deposition on Stenfilcon A and Narafilcon A Lenses
Description: Lens surface for narafilcon A and stenfilcon A is assessed. (Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe)
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Grade 0 | 64 | 62
  Grade 1 | 4 | 5
  Grade 2 | 0 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

7. Primary Outcome: Lens Surface - Wettability of Stenfilcon A and Narafilcon A Lenses
Description: Lens wettability for narafilcon A and stenfilcon A is assessed. (Grades 0-4, 0=normal, 1=trace, 2=mild, 3=moderate, 4=severe)
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Grade 0 | 55 | 59
  Grade 1 | 8 | 5
  Grade 2 | 4 | 4
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0

8. Primary Outcome: Lens Fit - Horizontal Centration of Stenfilcon A and Narafilcon A Lenses
Description: Horizontal centration assessed for narafilcon A and stenfilcon A lenses categorized as extremely nasal, slightly nasal, optimum, slightly temporal, extremely nasal.
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Extremely Nasal | 0 | 0
  Slightly Nasal | 0 | 0
  Optimum | 44 | 46
  Slightly Temporal | 24 | 22
  Extremely Temporal | 0 | 0

9. Primary Outcome: Lens Fit - Vertical Centration of Stenfilcon A and Narafilcon A Lenses
Description: Vertical centration assessed for narafilcon A and stenfilcon A lenses and graded as extremely nasal, slightly nasal, optimum, slightly temporal, extremely temporal.
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Extremely inferior | 0 | 0
  Slightly inferior | 11 | 12
  Optimum | 42 | 48
  Slightly superior | 15 | 8
  Extremely superior | 0 | 0

10. Primary Outcome: Lens Fit - Corneal Coverage of Stenfilcon A and Narafilcon A Lenses
Description: Corneal coverage will be assessed for narafilcon A and stenfilcon A and categorized as extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive.
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Extremely inadequate | 0 | 0
  Slightly inadequate | 4 | 2
  Optimum | 56 | 60
  Slighlty excessive | 8 | 6
  Extremely excessive | 0 | 0

11. Primary Outcome: Lens Movement
Description: Lens movement assessed for narafilcon A and senofilcon A lenses and categorized as extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive.
Time Frame: 1 week
Population: There were 2 participants excluded from the analysis for narafilcon A at 1 week due to protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Stenfilcon A | Narafilcon A
Number analyzed (Participants) | 68 | 65
Participants
  Extremely inadequate | 0 | 0
  Slightly inadequate | 3 | 5
  Optimum | 55 | 54
  Slightly excessive | 10 | 9
  Extremely excessive | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Description: Adverse events were collected during the study visit exams.
Groups:
- Stenfilcon A: Participants are randomized to wear stenfilcon A as the first or second lens pair for one week during the cross over study.
- Narafilcon A: Participants are randomized to wear narafilcon A as the first or second lens pair for one week during the cross over study.
Arm/Group | Stenfilcon A | Narafilcon A
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 2/70 | 6/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stenfilcon A (N=70) | Narafilcon A (N=70)
Non-ocular Non-Significant (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) — Common cold

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes